CLINICAL TRIAL: NCT04130048
Title: Assessment of Thrombus Stiffness Using Ultrasound Elastography in Venous Thrombo-embolism.
Brief Title: Thrombus Elastography in Venous Thrombo-Embolism.
Acronym: TEVTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: TEVTE ( 29BRC19. 101)
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-05

CONDITIONS: Venous Thromboembolism
Keywords: Elasticity Imaging Techniques; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound Elastography — Ultrasound elastography aims to assess the stiffness of a tissue, submitting it to an ultrasound impulse.

SUMMARY:
Venous Thrombo-Embolic Disease (VTED) is a serious and common ailment, defined by the growth of a clot - or thrombus - in a vein, and/or as the migration of this thrombus to a pulmonary artery. It represents the third cause of death after cardio-vascular disease and cancer, and encompass superficial, muscular and Deep Venous Thrombosis (DVT), and Pulmonary Embolisms (PE), which can be isolated or associated.

Ultrasound is today the most frequently used exam to diagnose DVT. However, it's unable to provide information on thrombus age or cause.

Elastography is an imaging technic which aims to analyse elastic properties of a tissue, by applying a mechanical impulse on it, and could be an interesting tool in thrombus exploration, and provide additional information.

DETAILED DESCRIPTION:
Proximal deep venous thrombosis of a lower limb was defined as any venous thrombosis involving the ilio-femoral and/or femoro-popliteal axes, with or without cava thrombosis or distal DVT.

A DVT was assumed provoked, as recommended by AFSSAPS (2009) and ACCP (2012), when there was a major transient risk factor (surgery, prolonged immobilization ≥3 days, lower limb fracture) in the last three months, or a persistent risk factor (Antiphospholipid syndrome, active cancer). In case of absence of at least one of these factors, DVT was considered unprovoked.

A DVT was supposed recent when there was no known DVT in the patient medical history.

The association with a Pulmonary Embolism was assessed by the presence of PE diagnosis in the medical report. It had to be diagnosed following the ESC guidelines, with a thoracic CT scan and/or a V/Q lung scan.

In this study, we analysed the shear wave's velocity (expressed in m/s).

Acquisitions were obtained during the venous ultrasound realised for the diagnosis of DVT. All measures were made on the same ultrasonic device, with the ShearWave module.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Suffering from a proximal DVT (DVT) of at least one lower limb.
* Thrombosis is assumed to be recent (no history of ipsilateral DVT).
* Non opposition obtained.

Exclusion Criteria:

* Patient suffering from an inferior vena cava thrombosis with no extension to ilio-femoral veins.
* Physical or cognitive inability to consent.
* Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient suffering from a proximal DVT (DVT) of at least one lower limb and admitted to the vascular medicine department of the Brest University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-12-14 (Estimated); Study Completion 2019-12-14 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Speed within the thrombus. | At VTE diagnostic (Day 0)
  Quantitative data, in meter per second.

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, Finistere, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.